CLINICAL TRIAL: NCT04153591
Title: Efficacy and Safety of Direct Oral Anticoagulants for the Treatment of Mural Thrombus
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 058.PHA.2019.D
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
To describe the prescribing patterns at Methodist Dallas Medical Center (MDMC) for the treatment of newly diagnosed mural thrombus and to determine the efficacy and safety of DOACs apixaban, dabigatran, and rivaroxaban in comparison to warfarin.

With limited treatment guideline consensus, minimal evidence to support the use of DOACs for Left Atrial Appendage (LAA) thrombus and Left Ventricular Thrombus (LVT), and a lack of evidence for the use of DOACs in aortic thrombus, further research is warranted to determine the role of DOACs in the treatment of various mural thrombi in comparison to warfarin.

DETAILED DESCRIPTION:
Retrospective chart review of MDMC patients from 4/1/2017 to 8/31/19 with newly diagnosed mural thrombus.

3.1. Study Methods

* Patients will be allocated into two groups: those who were prescribed DOACs upon discharge and those who were prescribed warfarin upon discharge
* Subgroup analyses will occur to evaluate the difference in efficacy and safety endpoints for patients into four categories including: those predisposed to mural thrombus by baseline risk factors (AFIB vs. ACS), location of the mural thrombus (atrial, ventricular, aortic), DOAC by agent (apixaban, rivaroxaban, dabigatran), and DOAC by scheduled dosing indication (AFIB vs. VTE).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. MHS patients with newly diagnosed mural thrombus from 4/1/2017 to 8/31/19 identified by International Classification of Diseases (ICD) codes: I23.6, I240, I513, I7409, I7411, I7419, I82210, I82229

Exclusion Criteria:

1. Age <18 years
2. Anticoagulant use at baseline (DOAC, LMWH, VKA)
3. Active cancer
4. Active bleeding
5. Pregnancy
6. Hospice or palliative care upon discharge
7. Warfarin that did not receive adequate bridging from parenteral anticoagulation
8. Non newly diagnosed mural thrombus

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospective chart review of MDMC patients from 4/1/2017 to 8/31/19 with newly diagnosed mural thrombus.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Efficacy of the direct oral anti-coagulants | from 4/1/2017 to 8/31/19
  Readmission for recurrent stroke or thromboembolic event within 90 days of initial hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Brown, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided